CLINICAL TRIAL: NCT03860285
Title: Objective and Perceived Quality Study in Patients Undergoing Elective Groin Hernia Surgery by the Abdominal Wall Surgery Unit of the Hospital Complex of Navarra
Brief Title: Objective and Perceived Quality Study in Patients Undergoing Elective Groin Hernia Surgery
Status: Suspended | Type: Observational
Why Stopped: Pending changes in recruitment
Sponsor: Hospital of Navarra (Other)
Responsible Party: Principal Investigator, Gorka Docio, General Surgeon, Senior, Hospital of Navarra
Other Study IDs: HNavarra
Record Dates: First submitted 2018-12-02; First posted 2019-03-01 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Inguinal Hernia; Quality of Life; Surgery; Survey
Keywords: inguinal hernia; quality of life; survey; surgery; pamplona; prospective; observational; cohorts
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Short form 36 quality of life survey — Prospective non-comparative observational study of cohorts
  Other Names: European Hernia Society Survey

SUMMARY:
This is a prospective non-comparative observational study of cohorts. Consists on offering surveys to every patient undergoing groin hernia surgery in our Abdominal Wall Surgery Unit, in Hospital of Navarra.

DETAILED DESCRIPTION:
HYPOTHESIS:

The objective and perceived quality data of the patients under study (adult patients undergoing scheduled inguinal hernia without complications) in Pamplona are within the international quality standards.

OBJECTIVES

Primary objective:

-Obtaining data of objective and perceived quality of patients undergoing elective groin hernia surgery in Pamplona durinag a year to compare them with international quality standards.

Secondary objectives:

* Obtaining data on duration of sick leave (temporary disability due to common contingency) associated with the referred procedures, as well as their possible complications.
* Assess the costs associated with the intervention and its possible complications.
* Raise options (if necessary and feasible) to improve the results exposed obtained by our service.

ELIGIBILITY:
Inclusion Criteria:

* Patients entering surgical waiting list during a year (from March 1st, 2018, to February 28th, 2019).
* Elective surgery.

Exclusion Criteria:

* Age below 16.
* Mental diseases.
* Patients not capable of understanding the study.
* Patients that reject entering the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing elective inguinal hernia surgery en Pamplona
Sampling Method: Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Obtaining objective and perceived quality of life | 4 years
  Obtaining data about objective and perceived quality of life of patients undergoing elective inguinal hernia surgery in Pamplona during a year to compare them with international quality standards

SECONDARY OUTCOMES:
Knowing patients' pain | 4 years
  Level of pain, before and after surgery
Registering hernia recurrence | 4 years
  Percentage of patients with hernia recurrence during study surveillance
Controlling presence or not of complications | 4 years
  Presence or not of postop complicationes
Knowing patient satisfaction | 4 years
  Grade of patient satisfaction with surgery result
Knowing duration of sick leave | 4 years
  How long is sick leave
Knowing waiting time for surgery | 4 years
  Patient waiting time until surgery date

CONTACTS AND LOCATIONS:
Overall Officials: Concepción Yárnoz-Irazabal, PhD, Study Director — Hospital de Navarra
Locations (1):
- Hospital de navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: Undecided